CLINICAL TRIAL: NCT06757088
Title: Effects of Combined Transcranial Direct Current Stimulation for Cerebral Cortex and Cerebellum on Postural Control in Elderly Population
Brief Title: Combined Effects of Transcranial Direct Current Stimulation on Postural Control in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Summaiya Ishtiaq/01899
Record Dates: First submitted 2024-10-08; First posted 2025-01-03 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Postural; Defect
Keywords: Posture; Old age; transcranial direct current

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- M1 Stimulation Group (MSG) (Active Comparator): For M1, the anodal electrode will be placed over M1 region while the cathodal electrode will be placed over the right contralateral supraorbital region.
  Interventions: Device: M1 Stimulation Group
- Cerebellar Stimulation Group (CbSG) (Other): For the CbSG, active anodal electrode will be placed over the cerebellum bilaterally about 1-2 cm below inion occipital protuberance, whereas the returning cathodal electrode will be placed on right buccinator muscle
  Interventions: Device: Cerebellar Stimulation Group (CbSG)
- M1 + cerebellar stimulation group (Experimental): In M1, the anodal electrode will be placed over the M1 region while the cathodal electrode will be placed over the right contralateral supraorbital region whereas simultaneously for the CbSG, active anodal electrode will be placed over the cerebellum bilaterally about 1-2 cm below inion occipital protuberance, whereas the returning cathodal electrode will be placed on right buccinator muscle
  Interventions: Combination Product: M1 + Cerebellar Stimulation Group
- Sham Stimulation group (SSG) (Sham Comparator): In Sham stimulation, Electrodes will be placed according to M1 Stimulation i.e., the anodal electrode will be placed over M1 region while the cathodal electrode will be placed over the right contralateral supraorbital region.
  Interventions: Device: Sham Stimulation Group

INTERVENTIONS:
Device: M1 Stimulation Group — For M1, the anodal electrode will be placed over M1 region while the cathodal electrode will be placed over the right contralateral supraorbital region.
  Arms: M1 Stimulation Group (MSG)
Device: Cerebellar Stimulation Group (CbSG) — For the Cerebellar Stimulation Group, active anodal electrode will be placed over the cerebellum bilaterally about 1-2 cm below the inion occipital protuberance, whereas the returning cathodal electrode will be placed on right buccinator muscle
  Arms: Cerebellar Stimulation Group (CbSG)
Combination Product: M1 + Cerebellar Stimulation Group — In M1, the anodal electrode will be placed over the M1 region while the cathodal electrode will be placed over the right contralateral supraorbital region whereas simultaneously for the CbSG, active anodal electrode will be placed over the cerebellum bilaterally about 1-2 cm below inion occipital protuberance, whereas the returning cathodal electrode will be placed on right buccinator muscle.
  Arms: M1 + cerebellar stimulation group
Device: Sham Stimulation Group — In Sham stimulation, Electrodes will be placed according to M1 Stimulation i.e., the anodal electrode will be placed over M1 region while the cathodal electrode will be placed over the right contralateral supraorbital region.
  Arms: Sham Stimulation group (SSG)

SUMMARY:
The current study aims to determine the effects of combination stimulation (M1 Cortex+ Cerebellum) along with balance training (X-box with Kinect) on postural control in elderly population and to compare the combined stimulation (M1+CbS) with individual motor cortex, cerebellar or sham stimulation.

DETAILED DESCRIPTION:
The current study has been designed to investigate the potential effects of short term transcranial direct current stimulation on motor cortex and cerebellum both simultaneously and to document any additional benefits over each individual stimulations (M1 cortex stimulation, cerebellar stimulation or sham stimulation). Patients will be receiving the transcranial direct current stimulation combined with non-immersive virtual reality using Xbox 360 with Kinect in each group.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Healthy elderly patients
* Age group of ≥ 60 years
* Fluent in reading and speaking Urdu language

Exclusion Criteria:

* Patients who have any congenital/Acquired walking or standing difficulty due to certain circumstances won't be included in the healthy adults group.
* Patients with Osteo-Arthritis (OA)
* Patients with cerebellar issues or issues such as vertigo with standing and walking etc.
* Individuals who had significant dysarthria or aphasia that might impair understanding of speech or verbal instruction
* Cognitive/communication impairment

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Berg balance scale (BBS) | 3 weeks
  Berg Balance Scale is considered gold standard for balance assessment. Patients are asked to complete 14 tasks, and each task is rated by an examiner on a 5-point scale ranging from 0 (cannot perform) to 4 (normal performance). Elements of the test are supposed to be representative of daily activities that require balance, including tasks such as sitting, standing, leaning over, and stepping. Some tasks are rated according to the quality of the performance of the task, whereas the time taken to complete the task is measured for other tasks. Overall scores can range from 0 (severely impaired balance) to 56 (excellent balance).
Timed Up and Go test (TUG) | 3 weeks
  The Timed Up and Go (TUG) test is a reliable, cost-effective, safe, and time-efficient way to evaluate overall functional mobility. The TUG has a high correlation with other proven tests that measure pure gait speed for longer lengths such as a 10-m walk.
Bestest Balance Evaluation-Systems Test (Bestest) | 3 weeks
  The Balance Evaluation Systems Test (BESTest) is a balance assessment that distinguishes 6 aspects of balance ability. Biomechanical constraints, limits of stability, anticipatory adjustments, postural responses, sensory orientation, and stability in gait. BESTest total score (ICC=0.98) and the BESTest sections (ICC between 0.85 and 0.96) have excellent intra-rater reliability. Inter-rater reliability for the total score was excellent (ICC=0.93) and, for the sections, it ranged between 0.71 and 0.94.
Twenty-five feet walk test (25FWT) | 3 weeks
  The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task. Administration time will vary depending upon the ability of the patient. Total administration time should be approximately 1-5 minutes. The T25-FW has high inter-rater and test-retest reliability and shows evidence of good concurrent validity.
Six-minute walk test (6MWT) | 3 weeks
  The 6-minute walk test (6MWT) is a sub-maximal exercise test used to assess aerobic capacity and endurance. It is a simple, non-invasive, low-cost and reproducible exercise test used to evaluate endurance during self-paced, submaximal walk by measuring the distance walked within 6 minutes (6MWD) along a flat, straight course with a hard surface. The 6-min walk had good test-retest reliability (88 < R < 94), particularly when a practice trial preceded the test trial.

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Nawaz Malik, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No